CLINICAL TRIAL: NCT04910932
Title: Effects of Breathing Exercises on Fear of COVID-19, Anxiety, Sleep and Quality of Life During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Collaborators: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Melih Zeren, Assist. Prof. Dr., Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bakircaymzeren04
Record Dates: First submitted 2021-06-01; First posted 2021-06-02 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercises group (Experimental): Breathing exercises will be applied via teleconference by a physiotherapist 1 day a week. Individuals will perform exercises by themselves at their homes on the remaining 6 days of the week. Exercise program will be applied for 4 weeks. Individuals will also be informed about COVID-19 for once at baseline.
  Interventions: Other: Breathing Exercises; Other: Information on COVID-19
- Control group (Other): Individuals will be informed about COVID-19 for once at baseline.
  Interventions: Other: Information on COVID-19

INTERVENTIONS:
Other: Breathing Exercises — Breathing exercises including diaphragmatic breathing, thoracic expansion and breathing control exercises
  Arms: Breathing Exercises group
Other: Information on COVID-19 — Information about COVID-19 based on the advices in "COVID-19 advice for the public" section of World Health Organization website.

SUMMARY:
It has been reported that in the first stages of the pandemic, a significant portion of the general population experienced psychological problems such as anxiety, depression and post-traumatic disorders. These problems persist today. A balanced diet, physical activity participation and relaxation techniques are recommended for preventing such problems. In studies conducted before the pandemic, it is reported that breathing exercises have positive effects on anxiety, sleep and quality of life in both patients and healthy individuals. Aim of this study is to investigate the effects of breathing exercises applied via teleconference on fear of COVID-19, anxiety, sleep and quality of life in healthy adult population.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study
* having a smart phone that can be used for teleconferencing purposes

Exclusion Criteria:

* have had COVID-19
* hospital admission for suspected COVID-19 in the past week
* having acute respiratory tract infection
* having any diagnosed chronic respiratory, cardiovascular, metabolic or neurological diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Fear of COVID-19 | Change from baseline at 2nd, 3rd and 4th week
  Fear of COVID-19 will be evaluated using The Fear of COVID-19 scale. The scale consists of seven items, each with a five-point Likert scale of options. The participant is instructed to choose an option that best represents their perception about the statement presented. Higher score indicates higher levels of fear.

SECONDARY OUTCOMES:
Anxiety | Change from baseline at 2nd, 3rd and 4th week
  Anxiety will be evaluated using Hamilton Anxiety Rating Scale. Scale measures the severity of a patient's anxiety, based on 14 parameters, including anxious mood, tension, fears, insomnia, somatic complaints and behavior. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Sleep quality | Change from baseline at 4th week
  Sleep quality will be evaluated using The Pittsburgh Sleep Quality Index. Questionnaire assesses sleep quality over a 1-month time interval. It consists of 19 individual items, creating 7 components that produce one global score. Each item is weighted on a 0-3 interval scale. The global score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Health-related quality of life | Change from baseline at 2nd, 3rd and 4th week
  Health-related quality of life will be evaluated using EQ-5D-3L. Questionnaire describes general health based on five distinct dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 Levels (indicating no problem, some or moderate problem and extreme problem).

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan University, Department of Physiotherapy and Rehabilitation, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Kepenek-Varol B, Zeren M, Dincer R, Erkaya S. Breathing and Relaxation Exercises Help Improving Fear of COVID-19, Anxiety, and Sleep Quality: A Randomized Controlled Trial. J Integr Complement Med. 2022 Jul;28(7):579-586. doi: 10.1089/jicm.2021.0381. Epub 2022 Apr 25. PMID 35467962